CLINICAL TRIAL: NCT00918840
Title: Antiretroviral-Sparing Concept: An Exploratory Phase II, Randomized, Single Blind Placebo-Controlled Study to Investigate the Effect of Therapeutic Immunization on the Quantity of HIV-Specific T Cell Precursors During Highly Active Antiretroviral Therapy Followed by Analytical Treatment Interruption
Brief Title: Antiretroviral-Sparing Concept With HIV-specific T Cell Precursors With High Proliferative Capacity (PHPC)
Acronym: PHPC-02
Status: Completed | Type: Observational
Sponsor: Genetic Immunity (Industry)
Collaborators: ViroStatics srl (Industry); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: PHPC-02; 2008-003765-11 (EudraCT Number)
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infection
Keywords: HIV; Vaccine; Immune Therapy; DermaVir; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — DermaVir; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells (PBMC) and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DermaVir + HAART: * Dosage: 0.4 mg DNA
  * Dosage form: 3.2 mL DNA/PEIm nanomedicine
  * Administration with 4 DermaPrep patches
  * Frequency: every 4 weeks
  * Duration: 8 weeks (3 DermaVir treatments)
  Interventions: Biological: DermaVir; Drug: HAART
- Placebo + HAART: * Dosage form: 3.2 mL Placebo
  * Administration with 4 DermaPrep patches
  * Frequency: every four weeks
  * Duration: 8 weeks (3 Placebo treatments)
  Interventions: Biological: Placebo; Drug: HAART

INTERVENTIONS:
Biological: DermaVir — DermaVir is a synthetic nanomedicine. The active pharmaceutical ingredient is a single plasmid DNA expressing 15 HIV proteins that assemble to HIV-like particles. DermaVir is topically administered with DermaPrep medical device to target the nanomedicine to Langerhans cells of the skin.These Langerhans cells migrate to the lymph node to induce cytotoxic T cells that can kill HIV-infected cells
  Other Names: LC002
  Groups: DermaVir + HAART
Biological: Placebo — Dextrose/glucose solution
  Other Names: LC002 Placebo
  Groups: Placebo + HAART
Drug: HAART — Three or more antiretroviral drugs that can fully suppress HIV RNA
  Other Names: Highly active antiretroviral therapy

SUMMARY:
PHPC-02 is a phase II, randomized, placebo-controlled trial designed to investigate whether therapeutic immunization during highly active antiretroviral therapy (HAART) induces elevations of HIV-specific T cell precursors with high proliferative capacity (PHPC) in HIV-1-infected individuals, and whether the quantity of PHPC correlates with the viral load set point following analytical treatment interruption (ATI). Subjects will be randomized to receive either DermaVir Patch (8 subjects per cohort) or DermaVir Patch Placebo (8 subjects per cohort) every four weeks for three applications while receiving maximally suppressive HAART. HAART will be discontinued at Week 9 for an ATI period of 20 weeks.

DETAILED DESCRIPTION:
16 subjects on maximally suppressive HAART were randomized to receive three doses of either DermaVir or Placebo immunotherapy.

Subjects receive three DermaVir/Placebo treatments over eight weeks (Weeks 0, 4 and 8) while receiving HAART. HAART is discontinued for a 20 week ATI.

Resumption of HAART during ATI is subjects experience:

* A confirmed CD4+ cell decrease by > 50%
* A confirmed CD4+ cell decrease to less than 350 counts/mL
* A confirmed VL increase > 300,000 copies
* Emergence of CDC AIDS related event(s)
* Signs or symptoms of clinically significant immunosuppression
* The subject or the subject's clinician wishes to restart HAART
* The subject becomes pregnant

ELIGIBILITY:
Main inclusion Criteria:

* HIV-1 infection
* On a non-hydroxyurea based HAART for at least one year
* Pre-HAART CD4 nadir > 250 cells/mm3
* Pre-HAART viral load > 5,000 copies/mL
* Undetectable viral load for the six month period preceding the study
* CD4 T-cell count >500 cells/mm3 for the six month period preceding the study

Main exclusion Criteria:

* No skin disease
* No hypersensitivity to adhesive tape or Tegaderm
* No history of keloid
* No history of vitiligo, melasma, skin cancer
* No tattoos or changes in pigment at the skin treatment sites
* No autoimmune diseases
* No hepatitis B, C coinfections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
HIV-specific memory T cells measured as PHPC count | 9 week
  DermaVir-induced PHPC count compared to Placebo

SECONDARY OUTCOMES:
HIV-1 RNA | weeks 16 and 20
  HIV-1 RNA set-point after analytical treatment interruption
CD4+ and CD8+ T cell counts | 20 weeks
Adverse Events | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renato Maserati, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia; Franco Lori, MD, Study Chair — ViroStatics srl
Locations (1):
- IRCCS Policlinico S. Matteo, Pavia, Italy

REFERENCES:
- [Background] Lisziewicz J, Toke ER. Nanomedicine applications towards the cure of HIV. Nanomedicine. 2013 Jan;9(1):28-38. doi: 10.1016/j.nano.2012.05.012. Epub 2012 May 30. PMID 22659241
- [Background] Lisziewicz J, Bakare N, Calarota SA, Banhegyi D, Szlavik J, Ujhelyi E, Toke ER, Molnar L, Lisziewicz Z, Autran B, Lori F. Single DermaVir immunization: dose-dependent expansion of precursor/memory T cells against all HIV antigens in HIV-1 infected individuals. PLoS One. 2012;7(5):e35416. doi: 10.1371/journal.pone.0035416. Epub 2012 May 9. PMID 22590502
- [Background] Lorincz O, Toke ER, Somogyi E, Horkay F, Chandran PL, Douglas JF, Szebeni J, Lisziewicz J. Structure and biological activity of pathogen-like synthetic nanomedicines. Nanomedicine. 2012 May;8(4):497-506. doi: 10.1016/j.nano.2011.07.013. Epub 2011 Aug 10. PMID 21839051
- [Background] Somogyi E, Xu J, Gudics A, Toth J, Kovacs AL, Lori F, Lisziewicz J. A plasmid DNA immunogen expressing fifteen protein antigens and complex virus-like particles (VLP+) mimicking naturally occurring HIV. Vaccine. 2011 Jan 17;29(4):744-53. doi: 10.1016/j.vaccine.2010.11.019. Epub 2010 Nov 23. PMID 21109034
- [Background] Calarota SA, Foli A, Maserati R, Baldanti F, Paolucci S, Young MA, Tsoukas CM, Lisziewicz J, Lori F. HIV-1-specific T cell precursors with high proliferative capacity correlate with low viremia and high CD4 counts in untreated individuals. J Immunol. 2008 May 1;180(9):5907-15. doi: 10.4049/jimmunol.180.9.5907. PMID 18424710
- [Background] Cristillo AD, Lisziewicz J, He L, Lori F, Galmin L, Trocio JN, Unangst T, Whitman L, Hudacik L, Bakare N, Whitney S, Restrepo S, Suschak J, Ferrari MG, Chung HK, Kalyanaraman VS, Markham P, Pal R. HIV-1 prophylactic vaccine comprised of topical DermaVir prime and protein boost elicits cellular immune responses and controls pathogenic R5 SHIV162P3. Virology. 2007 Sep 15;366(1):197-211. doi: 10.1016/j.virol.2007.04.012. Epub 2007 May 11. PMID 17499328
- [Background] Calarota SA, Weiner DB, Lori F, Lisziewicz J. Induction of HIV-specific memory T-cell responses by topical DermaVir vaccine. Vaccine. 2007 Apr 20;25(16):3070-4. doi: 10.1016/j.vaccine.2007.01.024. Epub 2007 Jan 22. PMID 17292518
- [Background] Lori F, Foli A, Lisziewicz J. Stopping HAART temporarily in the absence of virus rebound: exploring new HIV treatment options. Curr Opin HIV AIDS. 2007 Jan;2(1):14-20. doi: 10.1097/COH.0b013e328011aad6. PMID 19372860
- [Background] Xu JQ, Lori F, Lisziewicz J. CD4+ T cell-mediated presentation of non-infectious HIV-1 virion antigens to HIV-specific CD8+ T cells. Chin Med J (Engl). 2006 Oct 5;119(19):1629-38. PMID 17042976
- [Background] Lisziewicz J, Trocio J, Whitman L, Varga G, Xu J, Bakare N, Erbacher P, Fox C, Woodward R, Markham P, Arya S, Behr JP, Lori F. DermaVir: a novel topical vaccine for HIV/AIDS. J Invest Dermatol. 2005 Jan;124(1):160-9. doi: 10.1111/j.0022-202X.2004.23535.x. PMID 15654970
- [Background] Lisziewicz J, Trocio J, Xu J, Whitman L, Ryder A, Bakare N, Lewis MG, Wagner W, Pistorio A, Arya S, Lori F. Control of viral rebound through therapeutic immunization with DermaVir. AIDS. 2005 Jan 3;19(1):35-43. doi: 10.1097/00002030-200501030-00004. PMID 15627031
- [Background] Lori F, Kelly LM, Lisziewicz J. APC-targeted immunization for the treatment of HIV-1. Expert Rev Vaccines. 2004 Aug;3(4 Suppl):S189-98. doi: 10.1586/14760584.3.4.s189. PMID 15285717
- [Background] Foli A, Maserati R, Barasolo G, Castelli F, Tomasoni L, Migliorino M, Maggiolo F, Pan A, Paolucci S, Scudeller L, Tinelli C, D'Aquila R, Lisziewicz J, Lori F. Strategies to decrease viral load rebound, and prevent loss of CD4 and onset of resistance during structured treatment interruptions. Antivir Ther. 2004 Feb;9(1):123-32. PMID 15040544
- [Background] Lisziewicz J, Bakare N, Lori F. Therapeutic vaccination for future management of HIV/AIDS. Vaccine. 2003 Jan 30;21(7-8):620-3. doi: 10.1016/s0264-410x(02)00569-8. PMID 12531329
- See also: Genetic Immunity's homepage — http://www.geneticimmunity.com
- See also: Virostatics srl homepage — http://www.virostatics.com